CLINICAL TRIAL: NCT01293656
Title: Cross-sectional Study of Inflammatory Bowel Disease Severity and Treatment Patterns in Eastern Europe, Middle East, and North Africa. (P08166)
Brief Title: Study of Participants With Crohn's Disease and Ulcerative Colitis in Eastern Europe, Middle East, and North Africa (P08166)
Status: Withdrawn | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P08166
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CD and UC participants: All participants with CD or UC visiting their physician over a period of one year, newly and already diagnosed, regardless of treatment pattern.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — There is no study intervention. Participants will be treated locally per site standards.

SUMMARY:
This study is being done to assess the clinical course and treatment options for Crohn's Disease (CD) and ulcerative colitis (UC) in the populations of Eastern Europe, Middle East, and North Africa.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease or ulcerative colitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with CD or UC who visit the study sites in Eastern Europe, Middle East, and North Africa during the study period will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The number of participants with Crohn's Disease (CD) or ulcerative colitis (UC) who visit the participating sites. | 1 Year
The number of participants with different degrees of CD and UC severity. | 1 Year
Use rates of classes of drug therapy. | 1 Year
Number and types of surgical interventions. | 1 Year
Outcomes of surgical intervention. | 1 Year